CLINICAL TRIAL: NCT02552849
Title: Observational Study to Evaluate Disease Course and Outcomes in Patients Treated With Esbriet (Pirfenidone) for Idiopathic Pulmonary Fibrosis (IPF) in Canada
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29808
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Overall study: Specific treatment, dose, and treatment duration will be decided by the investigator independently of the participation of a patient in the study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This is a multi-center, non-interventional study to assess and describe course and outcomes in patients diagnosed with Idiopathic Pulmonary Fibrosis (IPF) who are treated with Esbriet (pirfenidone) in Canada, by measuring and reporting observed predicted forced vital capacity (FVC) change from baseline on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

* > or = 18 years of age
* Diagnosis of Idiopathic Pulmonary Fibrosis (IPF)
* Prescribed and/or currently taking Esbriet (pirfenidone) for the treatment of IPF

Exclusion Criteria:

* Hypersensitivity to Esbriet (pirfenidone)
* Concomitant use of fluvoxamine
* Severe hepatic impairment or end-stage liver disease
* Severe renal impairment or end-stage renal disease requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Idiopathic Pulmonary Fibrosis (IPF)
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2013-04-25 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Observed Predicted Forced Vital Capacity | Up to 4 years

SECONDARY OUTCOMES:
Proportion of Patients Not Taking Full Dose of Esbriet (pirfenidone) | Up to 4 years
Patient-Reported Outcome (PRO) Measure that Capture Quality of Life Using the A Tool Quality of Life Questionnaire (ATAQ-IPF) | Up to 4 years
Patient-Reported Outcome (PRO) Measure that Capture Quality of Life Using the Health-Related Quality of Life Questionnaire (HRQOL) | Up to 4 years
Patient-Reported Outcome (PRO) Measure that Capture Quality of Life Using the Work Productivity and Activity Impairment Questionnaire-General Health (WPAI-GH) | Up to 4 years
Patient-Reported Outcome (PRO) Measure that Capture Quality of Life Using the EuroQol-5 Dimension Questionnaire (EQ-5D) | Up to 4 years
Patient-Reported Outcome (PRO) Measure that Capture Quality of Life Using the St. George's Respiratory Questionnaire (SGRQ) | Up to 4 years
Progression-Free Survival (PFS) | Up to 4 years
Proportion of Patients Taking Full Dose of Esbriet (pirfenidone) | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- Canada (26):
  - South Health Campus/Alberta Health Services/ University of Calgary, Calgary, Alberta
  - Edmonton Respiratory Consultants & Edmonton Sleep Lab, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Synergy Respiratory Care, Sherwood Park, Alberta
  - Kelowna Respiratory and Allergy Cllinic, Kelowna, British Columbia
  - Mainra Rajesh R, Respirology, North Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital University of British Colambia Division of Hematology, Vancouver, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Clinique de pneumologie de Moncton Respiratory Clinic, Moncton, New Brunswick
  - Dr. Graham W. Bishop Clinic, Saint John, New Brunswick
  - Professional Medical Corporation, St. John's, Newfoundland and Labrador
  - St. Clare'S Mercy Hospital, St. John's, Newfoundland and Labrador
  - Burlington Lung Clinic, Burlington, Ontario
  - Firestone Institute for Respiratory Health, Hamilton, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario
  - Lawson Health Research Institute a joint venture of LHSC Research Inc and Lawson Research Institute, London, Ontario
  - Credit Valley Professional Building, Mississauga, Ontario
  - Oshawa Clinic, Oshawa, Ontario
  - Carling Respiratory Services, Ottawa, Ontario
  - Dr. Marc Newton Respirology, Owen Sound, Ontario
  - Toronto General Hospital; Investigational Pharmacy Services ENB - 217 (Pharmacy Receiving), Toronto, Ontario
  - Dr. Syed Anees Medicine Profession Corporation, Windsor, Ontario
  - Dr Anil Dhar Professional Medicine Corporation, Windsor, Ontario
  - Hopital Notre-Dame, Montreal, Quebec
  - Clinique de pneumologie et du sommeil de Lanaudiere, Saint-Charles-Borromée, Quebec